CLINICAL TRIAL: NCT00710398
Title: The Impact of Higher Dairy and Dietary Protein on the "Quality" of Hypoenergetic diet-and Exercise-induced Weight Loss in Pre-menopausal, Overweight and Obese Young Women
Brief Title: "Improving Diet, Exercise And Lifestyle (IDEAL) for Women" Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Dairy Farmers of Canada (Other); Dairy Management Inc. (Industry); Hamilton Health Sciences Corporation (Other)
Responsible Party: Dr. Stuart M. Phillips, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB 07-409
Record Dates: First submitted 2008-07-01; First posted 2008-07-04 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Overweight; Obesity
Keywords: Dairy Products; Dietary Protein; Body Composition; Fat mass loss; Lean mass gain; Pre-menopausal Women
MeSH Terms: conditions — Overweight; Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Experimental): A group consuming twice daily (post-exercise and in morning/afternoon) drinks containing no dairy protein or calcium. Daily protein intake (15% total kcals) should be from non-dairy sources (i.e. meat, egg, fish, chicken, wheat gluten).
  Interventions: Behavioral: Exercise - Aerobic and Resistance; Behavioral: Dietary - Caloric Restriction
- Dairy Protein (Experimental): A group consuming twice daily drinks (post-exercise and morning) containing 1% chocolate milk (in 1.5 cup servings = 3 cups/d). Daily protein intake is set at 15% total kcals with ~8% coming from dairy sources.
  Interventions: Behavioral: Exercise - Aerobic and Resistance; Behavioral: Dietary - Caloric Restriction
- High Dairy Protein (Experimental): A group consuming twice daily drinks of 1% artificially sweetened chocolate milk (in 1.5 cup servings = 3 cups/d). Their diet contains 30% protein (as opposed to only 15% in the Con and DairyPro groups) with at least 50% of that coming from dairy sources.
  Interventions: Behavioral: Exercise - Aerobic and Resistance; Behavioral: Dietary - Caloric Restriction

INTERVENTIONS:
Behavioral: Exercise - Aerobic and Resistance — Subjects will perform exercise (aerobic and resistance) 7d/wk and will exercise supervised 5d/wk. Exercise will be carried out to expend 250 kcals/day. Supervised resistance training sessions will take place 2 days/wk and aerobic exercise will take place every day. During the resistance exercise sessions, subjects will engage in a circuit weightlifting routine using guided motion machines. During the aerobic sessions, subjects may choose whatever exercise modality they like (e.g. walking on track or treadmill, biking, elliptical, etc.). Subjects will wear devices that measure energy expenditure to get a better idea of the intensity and duration needed to expend 250 kcals with their exercise machine/modality of choice.
Behavioral: Dietary - Caloric Restriction — Subjects will be counselled on their respective hypocaloric diets during the 16 wk period. Adherence to the prescribed diet will be assessed via collection of assigned food records (biweekly), frequent contact with subjects, and regular dietary counseling sessions. The daily dietary energy deficit will be 500 kcal per day based on the subjects' estimated daily caloric requirements (based on height, weight, age, sex), multiplied by a sedentary activity factor.
  Additionally, subjects will consume 2 drinks per day that will differ depending on their randomization allocation. Subjects in the Dairy Protein and High Dairy Protein group will be provided with dairy products (e.g. milk, cheese, yogurt) to consume on a weekly basis to help facilitate their prescribed dairy and dietary protein intake.

SUMMARY:
Diets all share the same principle: eat less energy than you need. This results in weight loss. However, the weight loss is usually a combination of a loss of body fat and muscle mass. Additionally, one's bones may begin to weaken, albeit very slowly, while on a diet, which could have serious long-term consequences. Thus, the investigators believe that the goal of any weight loss strategy should be to lose body fat and spare muscle. The investigators reasoning is two-fold. 1) Fat is not only stored under the skin, but also in and around the internal organs. When this occurs, the organ itself may not function properly. Losing fat mass is a very good thing from a health standpoint, since fat is not just a storage site for extra energy. Scientists have now shown that 'extra' body fat itself can actually secrete substances and when these substances get into your blood, they cause many problems and may even contribute to the development of diabetes. 2) Sparing muscle as an individual loses weight is very important. Muscle is a very 'metabolically active' tissue and is, by analogy, like the body's furnace. Muscle burns fuel from the food individuals eat and also from stored fuels, like fat. Hence, it's easy to see why you don't want to lose muscle because you'd be losing one of your body's best fat burners. More importantly, muscle is also a big storage site and furnace for blood sugar. In people with diabetes (elevated blood sugar), a big part of the problem is with their muscles - they simply do not take up and store or burn enough sugar. For these reasons, your goal should be to lose fat and preserve muscle while dieting.

There are many different diets to choose from (e.g. high protein, low carbohydrate, high fat, high fiber, etc.). A diet that has been shown to be quite successful, however, is one that is higher in protein (but not excessive). Thus, in this study, the investigators are proposing to test whether a higher protein (with dairy) and calcium diet promotes body fat loss and muscle mass retention. The investigators believe that a diet higher in protein (with an emphasis on dairy), but still within accepted healthy ranges, with higher dietary calcium may result in greater loss of body fat and retention of muscle than a diet with a conventional amount of protein and adequate calcium or a conventional amount of protein with little calcium (i.e. low dairy). Based on previous research, the investigators think that people with low calcium intakes to begin with would stand to benefit the most. There is also a good reason to think that the high protein/high calcium diet may result in greater reductions in blood cholesterol and blood sugar, both of which would reduce a person's risk for heart disease and diabetes.

The investigators will test this diet in premenopausal women who are overweight or obese. The investigators believe that this group is a good one to target for several reasons. First, women of this age who are overweight or obese are, if they continue to carry this excess weight, are at serious risk for developing chronic diseases such as heart disease, diabetes, and possibly cancer at an early age. Second, these women will often begin to gradually consume less dairy because many perceive dairy foods as fattening. Thus, if the investigators proposals are correct the investigators will hopefully be able to equip health professionals with a tried and tested, palatable, dietary strategy in a population segment who, because of their age, would benefit greatly were their disease risk to be reduced.

DETAILED DESCRIPTION:
Overweight to obese female subjects, who are habitually low dairy consumers and between the ages of 19-45 years will be recruited from the McMaster University student and staff population and from the surrounding Hamilton area. At study entry, all subjects will be asked to complete a standard screening questionnaire to document their medical history, current medication use, physical activity level, smoking habits, and alcohol consumption. Subjects will also complete a calcium food frequency questionnaire. Before randomization and study commencement, baseline measures will be done. These include: anthropometrics, fasting blood samples, fasting urine sample, resting energy expenditure measures (REE), muscle and adipose biopsies, cardiovascular measures (blood pressure, heart rate, blood vessel stiffness and arterial elasticity) body composition (dual-energy x-ray absorptiometry [DXA]), and a 7-day baseline food record analysis. Also, subjects' strength and fitness will be assessed (1 repetition maximum (RM) and submaximal Astrand Test evaluations). During the study, fasting blood samples will also be taken at weeks 4, 8, 12 and 16, DXA will also be done at weeks 8 and 16, validated Body Image questionnaires will be filled out again t weeks 8 and 16, and body weight will be recorded every week. All other measures will be repeated after 16 weeks (1RM, Astrand Test, biopsies, cardiovascular measures, REE). Magnetic Resonance Imaging (MRI) will be carried out on a smaller portion of subjects on a voluntary basis at weeks 0 and 16. Apon completion of the baseline testing, subjects will be randomly assigned to one of the three intervention groups.

Part of the intervention will be in the form of 2 daily chocolate drinks (a post-exercise drink plus one extra drink per day). Drink composition will differ depending on which group subjects are randomized to. Drinks will be made to look and taste similar. In terms of the daily diets, the DairyPro (middle/second) group will employ the same macronutrient distribution as the Control (first) group but half the protein will be derived from dairy sources, with subjects being asked to consume, on top of their supplemental chocolate drink, 2 yogurts (100 g each). In the control group, protein will be derived from sources other than dairy. In the HiDairyPro (third) group, dietary protein will be manipulated so as to comprise twice as much dietary energy versus the other two groups (i.e., 30% of energy intake versus 15%). Protein (half of their daily requirement) will be derived from dairy protein by asking subjects to consume, on top of their supplemental chocolate drink, 1 serving (250 ml) of 1% regular milk, 4 yogurts (100 g each) and 2 pieces of cheese (21 g each).

Overview of supplemental drink composition and diet composition by group:

1. Control (Con) - a group consuming twice daily drinks containing no dairy protein or calcium. Daily protein (15% total kcals) should be from non-dairy sources (i.e. meat, egg, fish, chicken, lentils, beans, wheat gluten).
2. Dairy Protein Group (DairyPro) - a group consuming twice daily drinks containing 1% chocolate milk and at least half of their daily protein (15% total kcals) intake from dairy sources.
3. High Dairy Protein Group (HiDairyPro) - a group consuming twice daily drinks containing 1% artificially sweetened chocolate milk along with a diet formulated to contain 30% (as opposed to only 15% in the Con and DairyPro groups) of their dietary energy from protein with at least half of that coming from dairy protein.

Subjects will meet with a study dietitian/nutritionist at the beginning and biweekly throughout the 16 weeks, and be provided with individual dietary counseling to reduce daily calories by 500 kcal/d. Subjects will be provided with template diet records, nutrition information sheets and macronutrient specific exchange lists to help with dietary compliance and to promote healthy food choices. The weight-reducing diets will have macronutrient and micronutrient profiles that are in accordance with the dietary regulations set forth by Canada's Food Guide and the dietary reference intakes (DRIs). The macronutrient profile of the 2 moderate protein groups (control and DairyPro) will be 15:30:55 (PRO:Fat:CHO), whereas the subjects in the High dairy protein group (HiDairyPro) will consume a profile of 30:30:40 (15% substitution of carbohydrate for protein). Subjects will consume all other food (aside from their designated drinks) in any manner they choose in accordance with the macronutrient profile of their respective randomization allocations. Adherence to the prescribed diet will be via collection of assigned biweekly food records, frequent contact with subjects, and regular dietary counseling sessions.

In addition, all subjects will be given a custom exercise prescription consisting of supervised resistance exercise and aerobic exercise. Intensity and duration of all exercise sessions will be monitored and energy expenditure quantified using portable, validated units that integrate accelerometry, heat flux and skin temperature. Exercise will take place in a supervised setting at McMaster University. Subjects will perform exercise 7d/wk and will exercise supervised 5d/wk (Mon - Fri). Resistance training sessions will take place 2x/week. During these sessions, subjects will engage in a circuit weightlifting routine using guided motion machines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pre-menopausal females
* Body Mass Index (BMI) between 27-40 kg/m2
* Low dairy consumption (~<500 mg/d Ca2+)
* Sedentary lifestyle (i.e., exercise less than once/week)
* Regular menstrual cycle

Exclusion Criteria:

* Allergy to dairy protein
* Lactose intolerance
* Vegan diet
* Pregnant
* Taking vitamin or mineral supplements
* Have a gastrointestinal disease or condition
* Recent orthopedic injury
* Diagnosed with heart, kidney, liver or pancreatic disease
* Smoker
* Alcohol consumption of more than 2 drinks/day

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-05 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Fat mass, lean mass, bone mass (BMD, BMC), total mass (measured via DXA scan) | Measured at weeks 0, 8 and 16

SECONDARY OUTCOMES:
Blood sample analyses (lipids) | Measured at weeks 0, 4, 8, 12 and 16
Muscle and adipose tissue biopsies | Measured at weeks 0 and 16
Food record macronutrient and micronutrient analyses (7-day at beginning and end, and 3-day throughout intervention) | Biweekly from weeks 0-16
Resting Energy Expenditure (metabolic cart determination). | Measured at weeks 0 and 16
Fitness and strength measures (modified Astrand Test and 1 RM test) | Measured at weeks 0 and 16
Blood sample analyses (Vitamin D [25OHD], PTH, A1c, glucose, insulin) | Measured at weeks 0 and 16
Magnetic Resonance Imaging (MRI) *strictly on a voluntary basis | Measured at weeks 0 and 16
Spot Urine Collection | Measured at weeks 0 and 16
Body Image (Assessed with a validated questionnaire) | Measured at weeks 0, 8 and 16
Cardiovascular Measures (Assessment of blood pressure, heart rate, blood vessel stiffness and arterial elasticity) | Measured at weeks 0 and 16

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M Phillips, Ph.D., Principal Investigator — Department of Kinesiology, McMaster University; Andrea R Josse, M.Sc., Study Director — Department of Kinesiology, McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Josse AR, Atkinson SA, Tarnopolsky MA, Phillips SM. Diets higher in dairy foods and dietary protein support bone health during diet- and exercise-induced weight loss in overweight and obese premenopausal women. J Clin Endocrinol Metab. 2012 Jan;97(1):251-60. doi: 10.1210/jc.2011-2165. Epub 2011 Nov 2. PMID 22049177
- [Derived] Josse AR, Atkinson SA, Tarnopolsky MA, Phillips SM. Increased consumption of dairy foods and protein during diet- and exercise-induced weight loss promotes fat mass loss and lean mass gain in overweight and obese premenopausal women. J Nutr. 2011 Sep;141(9):1626-34. doi: 10.3945/jn.111.141028. Epub 2011 Jul 20. PMID 21775530